CLINICAL TRIAL: NCT00751608
Title: A Randomized, Double-blind, Placebo-controlled Ascending Dose Study to Evaluate the Effect of APL180 on Endothelial Function in Patients With Familial Hypercholesterolemia
Brief Title: Effect of APL180 on Endothelial Function in Familial Hypercholesterolemia Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CAPL180A2207
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Familial Hypercholesterolemia
Keywords: Familial hypercholesterolemia, endothelial function, venous occlusion plethysmography, forearm blood flow, ApoAI-mimetic, endothelial dependent vasodilation
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: APL180
- 2 (Active Comparator)
  Interventions: Drug: APL180
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APL180
  Arms: 1
Drug: APL180
  Arms: 2
Drug: Placebo
  Arms: 3

SUMMARY:
This study will evaluate the effect of APL180 on endothelial function measured by forearm venous occlusion plethysmography in patients with familial hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed presence of familial hypercholesterolemia
* Women must be sterilized or post-menopausal

Exclusion Criteria:

* Smoking an average of greater than 10 cigarettes per day
* History of cardiac events
* Very low or high body weight
* Treatment with fibrates or niacin
* High blood triglyceride levels

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Change in forearm blood flow during each treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis Investigator Site